CLINICAL TRIAL: NCT02394301
Title: Efficacy of Novel Drug-combinations for Relief of Psoriasis (ENDURE)
Brief Title: Efficacy of Novel Drug-combinations for Relief of Psoriasis
Acronym: ENDURE
Status: Suspended | Type: Observational
Why Stopped: Poor enrollment
Sponsor: Medimix Specialty Pharmacy, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: Medimix Pharm-04
Record Dates: First submitted 2015-03-09; First posted 2015-03-20 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Psoriasis
Keywords: Efficacy of Novel Drug Combinations for Relief of Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: Yes

SUMMARY:
ENDURE is a prospective, observational study aimed to document clinical response and side effects associated with compounded psoriasis medications when prescribed as routine care. As a secondary initiative, this study will assess methotrexate systemic absorption and toxicity in patients prescribed a methotrexate-containing compounded formulation.

DETAILED DESCRIPTION:
In this prospective, observational study, change in psoriasis plaque appearance, per the Psoriasis Area Severity Index (PASI) tool, will be evaluated after using a topical psoriasis cream containing at least 3 of the following: corticosteroid, methotrexate, vitamin D3 or synthetic analog, retinoid acid, or urea, or a topical shampoo or spray containing a corticosteroid and vitamin D3 or synthetic analog. The change in quality of life will be assessed during all visits using the Skindex-16 assessment tool. In patients receiving a methotrexate-containing formulation, a sub-study will be available as an option, where laboratory values (methotrexate levels, complete blood count, liver function tests, etc.) will be obtained to confirm that methotrexate absorption is negligible.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Diagnosis of psoriasis vulgaris
* Being initiated on a topical compounded medication for psoriasis from Medimix Specialty Pharmacy containing at least 3 of the following ingredients as part of standard of care: corticosteroid, methotrexate, retinoic acid, vitamin D3 or synthetic analog, urea, AND/OR a shampoo/spray containing a corticosteroid and vitamin D3 or synthetic analog for the first time.

Exclusion Criteria:

* Pregnancy & nursing
* Active infectious disease
* Kidney abnormalities
* Blood deficiencies
* Alcohol consumption
* Immunodeficiency syndromes
* History of systemic psoriasis medications, including conventional DMARDs, oral retinoids, oral calcineurin inhibitors, TNF-inhibitors, and monoclonal antibodies within the past 120 days
* Current or planned use of concomitant psoriasis medications and/or phototherapy
* Any additional health conditions or concomitant use of other prescription/over-the-counter products that may confound the study results at the discretion of the study investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with psoriasis vulgaris that are prescribed a combination compounded topical psoriasis formulation.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-02; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change in Psoriasis Area Severity Index (PASI) Score | 12 Week Study [Baseline, 2, 4, 8, and 12 week evaluation]
  To evaluate the change in psoriasis plaque resolution, the PASI tool will be utilized. The psoriasis plaques will be evaluated by the overseeing study investigator as part of the normal evaluation of the area.

SECONDARY OUTCOMES:
Quality of Life | 12 Weeks [Baseline, 2, 4, 8, and 12 week evaluation]
  To assess change in quality of life, the Skindex-16 assessment tool will be used at all study visits.
Methotrexate absorption | 12 Weeks [Baseline, 4, 12 week evaluation]
  To assess changes in serum methotrexate concentration, methotrexate serum levels and other associated laboratory values (complete blood count, serum creatinine, alanine transaminase, aspartate aminotransferase, C-reactive protein, erythrocyte sedimentation rate, glucose, and insulin levels) will be monitored in patients that agree to participate in the sub-study who are prescribed a methotrexate-containing compounded psoriasis formulation (maximum 25 patients). This outcome measure is a composite.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin J Epstein, PharmD, Study Chair — Medimix Specialty Pharmacy
Locations (1):
- The Medimix Specialty Pharmacy, LLC, Jacksonville, Florida, United States

REFERENCES:
- [Background] Menter A, Griffiths CE. Current and future management of psoriasis. Lancet. 2007 Jul 21;370(9583):272-284. doi: 10.1016/S0140-6736(07)61129-5. PMID 17658398
- [Background] Tollefson MM, Crowson CS, McEvoy MT, Maradit Kremers H. Incidence of psoriasis in children: a population-based study. J Am Acad Dermatol. 2010 Jun;62(6):979-87. doi: 10.1016/j.jaad.2009.07.029. Epub 2009 Dec 5. PMID 19962785
- [Background] Choi J, Koo JY. Quality of life issues in psoriasis. J Am Acad Dermatol. 2003 Aug;49(2 Suppl):S57-61. doi: 10.1016/s0190-9622(03)01136-8. PMID 12894127
- [Background] Unaeze J, Nijsten T, Murphy A, Ravichandran C, Stern RS. Impact of psoriasis on health-related quality of life decreases over time: an 11-year prospective study. J Invest Dermatol. 2006 Jul;126(7):1480-9. doi: 10.1038/sj.jid.5700229. Epub 2006 Mar 30. PMID 16575395
- [Background] Krueger GG, Feldman SR, Camisa C, Duvic M, Elder JT, Gottlieb AB, Koo J, Krueger JG, Lebwohl M, Lowe N, Menter A, Morison WL, Prystowsky JH, Shupack JL, Taylor JR, Weinstein GD, Barton TL, Rolstad T, Day RM. Two considerations for patients with psoriasis and their clinicians: what defines mild, moderate, and severe psoriasis? What constitutes a clinically significant improvement when treating psoriasis? J Am Acad Dermatol. 2000 Aug;43(2 Pt 1):281-5. doi: 10.1067/mjd.2000.106374. PMID 10906652
- [Background] Armstrong AW, Robertson AD, Wu J, Schupp C, Lebwohl MG. Undertreatment, treatment trends, and treatment dissatisfaction among patients with psoriasis and psoriatic arthritis in the United States: findings from the National Psoriasis Foundation surveys, 2003-2011. JAMA Dermatol. 2013 Oct;149(10):1180-5. doi: 10.1001/jamadermatol.2013.5264. PMID 23945732